CLINICAL TRIAL: NCT01812798
Title: Disease Management: Canadian Peanut Thresholds Study
Brief Title: Canadian Peanut Thresholds Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McMaster University (Other)
Collaborators: AllerGen NCE Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 12LP3.7
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Peanut Allergy
Keywords: Peanut allergy; Threshold; Modelling; Risk assessment
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peanut (Active Comparator): Double Blind Placebo Controlled Food Challenge 5 gram peanut challenge
  17 doses of peanut will be administered. Dose will be increased every 20-30 minutes. All doses listed are in g of peanut flour.
  0.1 0.25 0.5 0.75
  1 2.5 5 10 25 50 100 250 500 750 1000 2500 5000
  Interventions: Other: Double Blind Placebo Controlled Food Challenge
- Placebo (Placebo Comparator): Double Blind Placebo Controlled Food Challenge (No peanut - placebo only)
  Interventions: Other: Double Blind Placebo Controlled Food Challenge

INTERVENTIONS:
Other: Double Blind Placebo Controlled Food Challenge — All participants will undergo Double Blind Placebo Controlled Food Challenge. Participants will be randomized to receive either Peanut on Day 1, Placebo on Day 2, or vice versa.
  For 'Peanut' arm, participants will be fed increasing doses of peanut until mild objective allergic reaction is observed.
  Doses will be increased every 20-30 minutes. All doses are listed in g peanut flour
  0.1 0.25 0.5 0.75
  1 2.5 5 10 25 50 100 250 500 750 1000 2500 5000
  For "Placebo" arm, participants will be fed increasing amounts of food matrix without peanut flour.

SUMMARY:
An important gap in the management of peanut allergy is that we do not know the threshold dose, below which most peanut allergic individuals will not react. There is likely a spectrum of reactivity to peanut where some individuals react to trace doses, whereas others are able to tolerate larger doses. The purpose of this study is to determine the minimum threshold dose needed to cause a mild objective reaction when peanuts are consumed by peanut-allergic individuals in a carefully controlled clinical setting. 30 peanut-allergic participants aged 7-65 years will undergo a two-day, double blind placebo controlled food challenge. Participants will be gradually fed increasing amounts of peanut, or placebo, until objective allergic symptoms are observed. Statistical modelling of individual threshold doses will be used to determine a population threshold dose, or a level of peanut to which 90% of the peanut-allergic population will not react. Knowledge of threshold doses at an individual and population level is valuable in that it provides critical information for the management of peanut allergy by individuals, their caregivers and health professionals, as well as knowledge of allergen risks to public health agencies and the food industry.

DETAILED DESCRIPTION:
Overview

This study protocol will be modeled on a consensus protocol developed with the input of clinical allergists and other allergy stakeholders to standardize threshold challenge studies [5-8]. As per protocol, 30 patients with a known or convincing history of peanut allergy will be recruited. After an initial screening visit to verify eligibility, all participants will undergo a two-day DBPCFC. Briefly, qualifying participants will be fed increasing amounts of peanut masked in a food matrix. On a different day, the participant will be fed the same amount of the food matrix without any peanut. Overall, the study will require three visits by participants: a screening day to determine if the prospective participants meet eligibility criteria, and two days for the DBPCFC.

Study Procedures

Screening Visit

Prospective participants will come to the Allergy Clinic at the McMaster University Medical Centre for a screening visit up to 6 months prior to the DBPCFC in order to confirm study eligibility. The informed consent form will be reviewed and signed at this time. The allergic status of these prospective participants will be characterized by patient history, skin prick test (SPT), and peanut-specific IgE, so that they can be related to the overall allergic population. Relevant history (all reactions related to peanut and any other foods, other allergic co-morbidities, other medical conditions, medications, family history, etc.) will be recorded. A physical examination will be performed including skin prick tests to peanut and the routine inhalant allergen panel. Blood work will be done as a baseline measure and analyzed as described below.

Skin Prick Test (SPT)

As a positive SPT is needed to qualify participants for the study, each prospective participant will have a SPT during the screening visit. SPTs will be judged and recorded based on the size of the wheal (raised welt around prick site) and flare (reddened area around wheal) as compared to the positive and negative control skin tests after 15-30 minutes [9]. A SPT is deemed positive by comparison to the negative control skin test. Skin test reaction wheals with diameters 3 mm greater than those of the negative saline control are considered positive. The diameter of the wheal and the diameter of the wheal and flare will be recorded. A record of the peanut SPT size will be kept via cellophane tape recording.

Blood draw

During the screening visit, a blood sample will be taken from prospective participants in order to test the in vitro peanut-specific IgE level. The amount of blood drawn will be dependent on the age and weight of the subject (see Appendix III). The blood will be separated so that the serum can be submitted for specific testing against peanut proteins. Testing for IgE to peanut requires only a few milliliters of serum. The remaining serum will be used to identify specific proteins in peanuts that bind IgE from each subject's serum and characterization of those peanut proteins. Serum samples will be coded to protect the identity of the subjects, stored at McMaster University Medical Centre, and used until supplies are exhausted.

Double Blind Placebo Controlled Food Challenge

Participants will come to the Allergy Clinic at McMaster University Medical Centre for the DBPCFC, which will take 2 days. Each visit will last a minimum of 4 hours with a minimum of one week between the food challenge visits. Oral food challenges will occur in a clinical setting allowing for prompt medical treatment if necessary during the protocol. Participants will be monitored by qualified medical personnel. An IV will be put in place prior to the start of the challenge. In the extremely unlikely event that the subject has a severe reaction during the challenge, a code cart or special emergency supplies including intubation equipment and defibrillator will be available and epinephrine and other medications will be administered according to the severity of reaction.

Each participant will be randomized to receive either peanut on Day 1 and placebo on Day 2 or vice versa. The randomization process and challenge materials are described in detail below. On the 'peanut' day, participants will be orally challenged with 17 doses of peanut masked in a suitable food matrix, such as applesauce or chocolate pudding. To ensure the establishment of a NOAEL, the starting dose will be 0.1mg, 50-30 times lower than what has previously been reported. The progression of dosing will follow a defined schedule up to 5000g. On a separate day, participants will be challenged with an equivalent series of placebo doses.

To start the challenge, each participant will be given a small amount of either peanut (masked in the challenge vehicle) starting at 0.1 mg or placebo. Doses will be given at 20-30 minute intervals and participants will be monitored continuously between doses. The dose of peanut will be increased following the progression above until:

1. One or more of the following objective findings are observed:

   1. Rash: erythema, morbilliform rash, urticarial, angioedema
   2. Ocular: conjunctival swelling, scleral edema, tearing
   3. Nasal: congestion, rhinorrhea, sneezing
   4. Gastrointestinal: vomiting, diarrhea
   5. Systemic: blood pressure drop by ≥ 20%
2. The final dose of peanut is reached
3. Physician's discretion

All subjective and objective symptoms will be fully recorded on the data collection forms. Vital signs (oxygen saturation, blood pressure, heart rate, respiratory rate) will be assessed before every dose, with every new subjective symptom reported, and when objective findings are observed. The challenge may be stopped at the discretion of the principal investigator if the participant cannot tolerate the subjective symptoms. Once objective reactive symptoms are observed, the challenge will immediately be stopped and the participant will receive appropriate medication which may include epinephrine, antihistamine, or steroids to manage the reaction. Participants will be observed for a minimum of 2 hours after an allergic reaction has occurred to ensure that it has been adequately treated and resolved.

ELIGIBILITY:
Inclusion Criteria:

1. Children and adults between 7-65 years of age.
2. Demonstrated history of peanut allergy based on medical history, positive skin prick test, and peanut-specific IgE CAP-FEIA test. Participants will be confirmed to have peanut allergy based on a history of significant clinical symptoms within 60 minutes of the ingestion of peanut, the presence of specific IgE to peanut (a positive skin prick test to peanut, defined as a wheal 3 mm larger than that of the saline control, and a positive in vitro peanut-specific IgE (CAP-FEIA) test value >0.35 IU/mL.
3. Ability to discontinue all prescribed and over the counter allergy-related medications for suitable withdrawal periods before starting the challenge trial. See Appendix I for specifications.

Exclusion Criteria:

1. Previous desensitization treatment to peanut
2. Allergies to any component of the oral challenge matrix
3. Unstable allergic conditions such as uncontrolled asthma or chronic urticaria
4. Any clinically significant disease/chronic medical condition which may interfere with study evaluations

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-05; Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Peanut threshold dose | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Susan Waserman, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada